CLINICAL TRIAL: NCT00465231
Title: Preventive Analgesia in Labour:A Randomised, Placebo-Controlled Study in Multiparas Undergoing Induction of Labour
Brief Title: Preventive Analgesia in Multiparas Undergoing Induction of Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Dr. Jose Carvalho, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07-01; 06-0230-A
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Pain
Keywords: Induction of labour; Bupivacaine consumption; Prevention
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Epidural
  Interventions: Drug: bupivacaine, fentanyl
- 2 (Placebo Comparator): Epidural - saline solution
  Interventions: Drug: preservative free saline

INTERVENTIONS:
Drug: bupivacaine, fentanyl — 10mL of 0.0625% of bupivacaine plus fentanyl 2 mcg/ml
  Arms: 1
Drug: preservative free saline — 10mL saline solution
  Arms: 2

SUMMARY:
Our study is about providing a better birthing experience by placing and initiating epidural for labour pain before the contractions start. This concept of prevention of pain before its onset is known as preventive - or preemptive -pain management and is well known in surgical and anaesthetic practice. We believe that the use of preventive epidural analgesia will improve the quality of labour epidurals, increase maternal satisfaction and reduce the stress response to labour and delivery.

DETAILED DESCRIPTION:
Labour induces a well-documented stress response in both mother and fetus. Pain, anxiety and stress associated with labour result in the activation of the sympathetic nervous system, which increases plasma catecholamine concentrations with a resultant increase in cardiac output, peripheral vascular resistance and eventually, reduction in utero-placental perfusion. One aspect that has not been addressed in the literature is the role of preventive analgesia in labour. We believe that the use of preventive epidural analgesia will improve the quality of labour pain, increase maternal satisfaction and reduce the stress response in labour.

The multiparous parturients that are scheduled for elective inductions of labour will be offered preventive epidural analgesia. Upon placing the epidural, patients will receive, in a double blind fashion, one of two possible epidural drug regimens, which are a saline placebo or 0.0625% bupivacaine with 2 micrograms of fentanyl per millilitre. The patient then undergoes routine induction and management of labour. At any point after induction of labour, patients in either group can request analgesia. Upon request for analgesia the standard epidural loading dose and infusion with PCEA is initiated. The primary outcome will be the success of analgesia (Verbal Analogue Scale of 3 or less) during the first stage of labor, from first request of epidural analgesia to full dilatation.

ELIGIBILITY:
Inclusion Criteria:

* Multiparous patients who had previous vaginal delivery, undergoing induction of labour
* Singleton Pregnancy

Exclusion Criteria:

* Morbid Obesity
* Patients who have received cortisol, opioids or sedatives within the last 24 hours

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Pain scores (VAS) remain 3 or less | throughout the first stage of labor

SECONDARY OUTCOMES:
Bupivacaine consumption | during labour
Urinary creatinine to cortisol ratio | during labour
Neonatal outcome | at delivery
Obstetric outcome | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD PhD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada